CLINICAL TRIAL: NCT06402019
Title: Repeated Dexmedetomidine Infusion is a Two-shot Weapon for Pain and Pain-induced Mood Disorders in Chronic Pain Patients
Brief Title: Dexmedetomidine Infusion Impact on Chronic Pain Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Salsabil Sayed Abdelkader, Clinical lecturer at Department of Anesthesia, Pain & ICU, Faculty of Medicine, Benha University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RC.9.3.2024
Record Dates: First submitted 2024-04-13; First posted 2024-05-07 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain | interventions — Dexmedetomidine; Saline Solution

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Active Comparator)
  Interventions: Drug: Dexmedetomidine in 0.9 % NaCl 20 Mcg/5 mL (4 Mcg/mL) INTRAVEN SYRINGE (ML)
- Control Group (Placebo Comparator)
  Interventions: Drug: normal saline

INTERVENTIONS:
Drug: Dexmedetomidine in 0.9 % NaCl 20 Mcg/5 mL (4 Mcg/mL) INTRAVEN SYRINGE (ML) — Group went under multiple sessions of Dexmedetomidine infusion for 10 sessions; The infusion was provided under non-invasive monitoring for heart rate (HR) and mean arterial pressure (MAP). The infusion rate was adjusted to maintain HR in range of 60-80 beats/min and MAP in range of 65-75 mmHg.
  Arms: Intervention Group
Drug: normal saline — Group went under multiple sessions of normal saline injection.
  Arms: Control Group

SUMMARY:
Chronic pain (CP) was defined as pain experienced daily or on most days and induced restriction of at least one activity. CP is one of the commonest complaints confronted in outpatient clinics and constitutes a challenge for all medical provisions. CP is a multifaceted condition; postoperative CP is frequently encountered in clinical practice and may be of debilitating severity leading to worse quality of life (QOL) especially CP with a neuropathic component as post-mastectomy pain syndrome and post-amputation pain and chronic post-sternotomy pain that seriously impacts patients' QOL and affects patient recovery till 12 months after cardiac surgery. Chronic musculoskeletal pain as defined by the International Pain Association is the persistent or recurrent pain involving spine, bones, joints, and/or musculo-soft tissue.

Chronic pain was considered as a long-lasting stressor that might induce disordered mood varying between depression and anxiety with consequent challenge of this combination on treatment outcomes and consumption of health resources. This necessitated psychological screening of CP patient to identify and manage patients with disordered mood to improve CP treatment outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients with multiple-level spinal canal stenosis who refused surgical management.

Exclusion Criteria:

* Patients with other causes for CP;
* maintained on opioid analgesia;
* had cardiac lesions;
* maintained on antihypertensive therapy;
* hepatic impairment;
* Patients can't attend the clinic to complete the course of Dexmedetomidine infusion sessions.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-09-22 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
The extent of reduction of consumed analgesics | 6 months
  Necessity of Dexmedetomidine infusion as management procedure to the chronic pain patients

CONTACTS AND LOCATIONS:
Locations (1):
- Benha university, Banhā, Qalyoubia, Egypt